CLINICAL TRIAL: NCT07263776
Title: Efficacy and Safety of Interleukin-6 Receptor Inhibitor Combined With Endovascular Treatment in Patients With Acute Anterior Circulation Large Vessel Occlusion Stroke: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial-2 (IRIS-2)
Brief Title: Efficacy and Safety of Interleukin-6 Receptor Inhibitor Combined With Endovascular Treatment in Patients With Acute Anterior Circulation Large Vessel Occlusion Stroke -2
Acronym: IRIS-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRIS-2
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Interleukin-6 Receptor Inhibitor; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab group (Experimental): Endovascular treatment combined 240 mg tocilizumab injection once.
  Interventions: Drug: Tocilizumab
- Placebo group (Placebo Comparator): Endovascular treatment combined equivalent volume of placebo once.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — 240 mg of tocilizumab injection will be diluted in 0.9% NaCl solution to prepare a total solution volume of 100 mL. The solution will be administered via intravenous infusion immediately after randomization, and no later than 30 minutes, with an infusion duration of more than 1 hour.
  Arms: Tocilizumab group
Drug: Placebo — An equivalent volume of placebo will be diluted in 0.9% NaCl solution to prepare a total solution volume of 100 mL. The solution will be administered via intravenous infusion immediately after randomization, and no later than 30 minutes, with an infusion duration of more than 1 hour.
  Arms: Placebo group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial. Investigators aim to assess the efficacy and safety of interleukin-6 receptor inhibitor combined with endovascular treatment in patients with acute anterior circulation large vessel occlusion stroke.

DETAILED DESCRIPTION:
The study population are patients with acute anterior circulation large vessel occlusion stroke and planned to undergo endovascular treatment. All participants are randomly assigned in a 1:1 ratio to the tocilizumab group or the placebo group. In tocilizumab group, participants will receive tocilizumab combined endovascular treatment. And in placebo group, participants will receive placebo combined endovascular treatment. All participants will be visited immediately postoperatively, at 24 hours, 7 days, and 90 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater, male or female;
2. Acute ischemic stroke caused by occlusion of intracranial segment of the internal carotid artery, middle cerebral artery M1 or proximal/dominant M2 segment;
3. Decided to undergo emergency endovascular treatment;
4. Time from stroke onset to arterial puncture within 24 hours;
5. National Institutes of Health Stroke Scale (NIHSS) score ≥ 6;
6. Signed informed consent from the patients or the legally authorized representatives.

Exclusion Criteria:

1. Intracerebral hemorrhage, epidural hematoma, subdural hematoma, intraventricular hemorrhage, or subarachnoid hemorrhage;
2. Pre-stroke modified Rankin scale (mRS) score >1;
3. Known allergy to tocilizumab or excipients;
4. Known allergy to iodinated contrast agents;
5. Anticipated difficulty in completing endovascular treatment due to vascular tortuosity;
6. History of congenital or acquired bleeding disorders, coagulation factor deficiency diseases, or thrombocytopenic diseases;
7. Systolic blood pressure ≥180mmHg or diastolic blood pressure ≥110mmHg despite blood pressure control;
8. Neutrophils <2×109 /L;
9. Platelets <100×109 /L;
10. Blood glucose <2.8mmol/L (50 mg/dL) or >22.2mmol/L (400 mg/dL);
11. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >2 times the upper limit of normal;
12. Known recent or current serum creatinine >2 times the upper limit of normal or estimated glomerular filtration rate (eGFR) <60 mL/min;
13. Pregnant, lactating, or planning pregnancy within 90 days;
14. Severe mental disorders or inability to comply with informed consent and follow-up requirements due to dementia;
15. Concurrent malignant tumors or severe systemic diseases with expected survival of less than 90 days;
16. Presence of autoimmune diseases or use of immunosuppressive drugs;
17. Systemic infectious diseases;
18. Participation in another interventional clinical study within 30 days before randomization or currently participating in another interventional clinical study;
19. Considered by the investigator to have other conditions that might affect compliance or preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score at 90 days | 90 days
  The mRS ranges from 0 to 6, with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Proportion of patients with mRS score 0-2 at 90 days | 90 days
Proportion of patients with mRS score 0-1 at 90 days | 90 days
National Institutes of Health Stroke Scale (NIHSS) score at 7 days or at early discharge | 7 days or at early discharge
  The NIHSS ranges from 0 to 42, with higher scores indicating worse outcomes.
Infarct volume at 24 hours | 24 hours
EuroQol Five-Dimension Five-Level Questionnaire (EQ-5D-5L) at 90 days | 90 days
  The EQ-5D-5L includes 5 dimensions: mobility, self-care, usual activities,pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scoresindicating worse quality of life.
Proportion of Barthel Index (BI) 95-100 at 90 days | 90 days
Incidence of symptomatic intracerebral hemorrhage within 24 hours | 24 hours
Incidence of any intracerebral hemorrhage within 24 hours | 24 hours
Proportion of patients with pneumonia at 7 days or at early discharge | 7 days or at early discharge
Mortality at 90 days | 90 days

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Si Country People's Hospital, Suzhou, Anhui
  - Lingshan County People's Hospital, Qinzhou, Guangxi
  - The second Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Yutian Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The People's Hospital of Anyang, Anyang, Henan
  - Jun County People's Hospital, Hebi, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tianyou Hospital Affliated to Wuhan University of Science &Technology, Wuhan, Hubei
  - Xiangyang No.1 People's hospital, Xiangyang, Hubei
  - Xing'an league People's Hospital, Xing’an, Inner Mongolia
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - People's Hospital of Dongying, Dongying, Shandong
  - Linshu Country People's Hospital, Linyi, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Huangdao District Hospital of Traditional Chinese Medicine, Qingdao, Shandong
  - Yiyuan Country People's Hospital, Zibo, Shandong
  - Shanxi Medical University First Hospital, Taiyuan, Shanxi
  - The People's Hospital of Xianyang, Xianyang, Shanxi
  - Daliuta Experimental District People's Hospital of Shenmu City, Yulin, Shanxi
  - Zhongxiang Traditional Chinese Medical Hospital, Zhongxiang, Wuhan
  - Xuanwu Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Related data will be shared if full study protocol and statistical analysis plan are provided with reasonable design.